CLINICAL TRIAL: NCT01684774
Title: Comparison Between Ultrasound-guided and Landmark-guided Ankle Blocks
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0070-12-HYMC
Record Dates: First submitted 2012-09-10; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2012-09

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- I. USG: Patients receiving Ultrasound-guided Ankle Block
  Interventions: Drug: Bupivacaine
- II. ALG: Patients receiving Anatomic Landmark-guided Ankle Block
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine

SUMMARY:
The investigators will be comparing ultrasound-guided (USG) ankle block and anatomic landmark-guided (ALG) ankle block to determine which of these procedures is better in surgical anesthesia and in postoperative pain relief.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthopedic foot operation with osteotomy

Exclusion Criteria:

* Skin infection near block injection site
* Allergy to local anesthetics
* Coagulopathy with INR >1.4.
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ASA I-III (American Society of Anesthesiologists classification) patients undergoing orthopedic foot operation with osteotomy
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Anesthesia Sufficient | Thirty minutes
  Sufficiency of surgical anesthesia will be determined by the presence of a complete sensory or motor block. If general anesthesia needs to be added to achieve operative analgesia, the surgical block will not be deemed sufficient.
Post-operative Pain Relief | Twenty-four hours
  Intensity of post-operative pain will be measured by a numerical scale from 0-10 by the patient

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel